CLINICAL TRIAL: NCT02065518
Title: Electromyostimulation and Strength Walking for Knee Injuries
Acronym: KI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); Malcolm Grow Medical Clinics and Surgery Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HU0001-10-1-TS04; TSNRP Grant HU0001-10-1-TS04 (Other Grant/Funding Number: TSNRP)
Record Dates: First submitted 2014-02-12; First posted 2014-02-19 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-10

CONDITIONS: Knee Injury
Keywords: Muscle strength; Electrical muscle stimulation; Strength training
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard Rehabilitation Protocol (SRP) (Active Comparator): All participants will receive the current standard of care, the physical therapy rehabilitation protocol for knee injuries at the WRNMMC and MGMCSC sites. This program includes treatment supervised by a physical therapist at the physical therapy clinics.
  Interventions: Behavioral: Standard Rehabilitation Protocol
- NMES w/ SRP (Experimental): In addition to the standard rehabilitation protocol, two treatment groups will receive a portable lightweight device (300PV unit) that provides clearly defined electrical stimuli. NMES training will consist of performing four 30-minute stimulation sessions per week for 12 weeks; each 30-minute session will entail 15 minutes/leg with 15 contractions per leg. Each contraction will be elicited by an electrical impulse (300PV) generated by a battery-operated device (EMPI, St. Paul, MN).
  Interventions: Device: NMES; Behavioral: Standard Rehabilitation Protocol
- Strength Walking w/ SRP (Experimental): The Strength Walking groups will participate in a Home-Based Pedometer-Driven Walking Program. All participants in this group will be given a pedometer to monitor their daily steps and, at week 7, a weighted exercise vest to begin the strengthening component. In addition to the standard WRNMMC rehabilitation protocol, a series of 10-minute lessons focused on increasing physical activity through lifestyle education and the use of a pedometer as a motivational tool and personal fitness tracker will be incorporated into their testing sessions for the first 6 weeks. At week 7, participants will be given a weighted vest to begin the strengthening component.
  Interventions: Behavioral: Strength Walking; Behavioral: Standard Rehabilitation Protocol
- NMES/Strength Walking w/ SRP (Experimental): In addition to the standard rehabilitation protocol, one group will receive NMES training and will participate in a Home-Based Pedometer-Driven Walking Program. This group will follow the protocol for both the NMES training and Strength Walking.
  Interventions: Device: NMES; Behavioral: Strength Walking; Behavioral: Standard Rehabilitation Protocol

INTERVENTIONS:
Device: NMES — Participants will train at 15-20% of maximal voluntary contraction (MVC) during weeks 1-3, 21-30% of MVC during weeks 3-6 and 31-40% of MVC during weeks 6-9, 41-50% of MVC during weeks 9-12, then sustain 50% of MVC during weeks 12-18. Incremental increases will be made at the 3, 6, 9, and 12-week clinic visits.
  Other Names: EMPI 300PV neuromuscular stimulator
  Arms: NMES w/ SRP; NMES/Strength Walking w/ SRP
Behavioral: Strength Walking — Strength Walking participants will maintain a daily training log. Pedometer readings will form the basis for setting activity goals. Initial step goals will be 10% above the average 3-day pedometer step count taken at baseline, with a 10% increase every other week, and then a gradual increase when 30% above the baseline step count has been achieved. At week 7, participants will be given a weighted vest to begin the strengthening component. Participants will be instructed to wear the vest during their 30-minute walk, 3 to 4 days a week. The beginning weight load for the vest will be calculated using 2% of baseline body weight and it will be increased by that same amount every week thereafter until the end of the 12 weeks.
  Arms: NMES/Strength Walking w/ SRP; Strength Walking w/ SRP
Behavioral: Standard Rehabilitation Protocol — All participants will receive the current standard of care at the 2 military sites (Walter Reed National Military Medical Center (WRNMMC) and Malcolm Grow Medical Clinics and Surgery Center (MGMCSC)) of the physical therapy rehabilitation protocol for knee injuries. This program includes treatment with a physical therapist at WRNMMC and MGMCSC physical therapy clinic.

SUMMARY:
The purpose of this project is to compare three treatment regimens for knee injury to the standard rehabilitation protocol: 1) NMES, 2) graduated strength walking (via a weighted vest), and 3) NMES combined with graduated strength walking. Each treatment arm will be supplemented by the standard of care and compared to a group who receive the standard rehabilitation only.

The Study will compare the effects of NMES, Strength Walking and combined NMES/ Strength Walking on strength, mobility, symptomatology, and Quality of Life (QOL) in military members with knee injury to a standard rehabilitation protocol program only. All groups will participate in standard rehabilitation protocol. The groups will be assessed over 18 weeks to compare main and interactive effects over time.

DETAILED DESCRIPTION:
The prevalence of knee injuries has shown a striking increase of >24% over the last 5 years, affecting work performance, limiting mobility, and impacting military deployment health. This increase reflects the current high op-tempo and frequent deployments of a nation at war including activities related to military operations, physical fitness, and demanding training. We have shown that neuromuscular electrical stimulation (NMES) improves quadriceps muscle strength. We have also shown that a pedometer-based protocol improves fitness. The overall objective of this project is to compare three treatment regimens for knee injury to the standard rehabilitation protocol as potential treatments for improving strength, work efficiency, and mobility in active duty military personnel with a knee injury. Our central hypothesis is that the combination of NMES and walking while wearing a weighted vest will demonstrate greater improvements in muscle strength, work efficiency, and mobility, as compared to the usual care alone. The rationale is that NMES combined with graduated strength walking could produce marked improvements in muscle strength and thereby enhance work performance, readiness and fitness, decrease physical symptoms and faster return to duty. NMES and graduated strength walking, simulate the current uniform in the theatre of operation (body armor).The specific aims are to compare the effectiveness of three treatment regimens to the usual care in improving: (1) muscle strength, (2) work efficiency, (3) mobility, (4) symptoms/pain, and (5) quality of life. After baseline testing, we propose to randomly assign male and female subjects (n=132) ages 18 to 50 years with a knee injury to one of 4 groups: 1) NMES, 2) strength walking, 3) NMES and strength walking, or 4) usual care. All groups will receive 12-weeks of the intervention and 6-weeks of follow-up. Generalized estimating equation (GEE) methods will be used to build regression models for statistical analysis of longitudinal data. If the interventions are effective with respect to parameters of strength, mobility, work performance, and symptoms, recommendations for future treatments can be made. This is hugely important, given the rising rate of knee injuries and the possibility that provider-managed care would be critical for assisting our warriors in a rapid recovery and return to duty.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of knee injury (internal derangement of the knee with new effusion, including knee sprain or strains, meniscal tear, cruciate ligamentous tear, and chondral flap or injury);
* A diagnosis of knee pain that is anterior knee pain, overuse pain, patella-femoral pain, and chronic pain (less than 6 months) associated with overuse syndromes which negatively impacts performance by (a) pain in 1 or both knees on most days of the month; b) self reported difficulty performing at least one or more tasks due to pain: stair climbing, rising from a chair, walking or running a quarter mile, repetitive movements such as kneeling or squatting or stooping, pain that inhibits job performance and daily activities;
* Military service member at the time of injury (active duty military and Reserve/ National Guard in active duty status);
* Age ≥18 and ≤50 years;
* Ability to provide freely given informed consent.

Exclusion Criteria:

* Fracture or injury to external knee structures such that knee extension or flexion is impaired;
* Evidence of a fracture on radiographs or clinical evidence of unstable tendon tear/rupture;
* A significant co-morbid medical condition (such as severe hypertension or neurological disorder in which NMES strength training or unsupervised exercise is contraindicated and would pose a safety threat or impair ability to participate;
* Inability or unwillingness to participate in a walking or strengthening program;
* Inability to speak and/or read English;
* Reduced sensory perception in the lower extremities;
* Inability to walk on a treadmill without an assistive device;
* Vision impairment, where participant is classified as legally blind;
* Unwillingness to accept random assignment;
* Pregnancy;
* A score of 23 or greater on the Center for Epidemiological Studies- Depression scale (CES-D);
* If the person has a demand type implanted pacemaker or defibrillator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Talbot, PhD, RN, Principal Investigator — University of Tennessee Health Sciences Center
Locations (2):
- United States (2):
  - Malcolm Grow Medical Clinics and Surgery Center, Andrews Air Force Base, Maryland
  - Walter Reed National Military Medical Cener, Bethesda, Maryland

REFERENCES:
- [Background] Talbot LA. (2016). Electromyostimulation and Strength Walking for Knee Injuries: Nurse Managed Care. 19 p, NTIS Report No.: PB2017102173.
- [Result] Talbot LA, Brede E, Price MN, Zuber PD, Metter EJ. Self-Managed Strength Training for Active Duty Military With a Knee Injury: A Randomized Controlled Pilot Trial. Mil Med. 2019 Jul 1;184(7-8):e174-e183. doi: 10.1093/milmed/usy347. PMID 30690578
- [Derived] Talbot LA, Brede E, Price M, Metter EJ. Health-related quality of life in active duty military: A secondary data analysis of two randomized controlled trials. Nurs Outlook. 2017 Sep-Oct;65(5S):S53-S60. doi: 10.1016/j.outlook.2017.07.010. Epub 2017 Jul 25. PMID 28830632

RESULTS

PARTICIPANT FLOW:
Groups:
- NMES w/ SRP: NMES (EMPI 300PV stimulator) plus SRP: NMES training consisted of four 30-minute stimulation sessions per week for 12 weeks; each 30-minute session entails 15 minutes/leg with 15 contractions per leg.
  Weeks 1-3: 15-20% of maximal voluntary contraction (MVC); Weeks 3-6: 20-30% of MVC; Weeks 6-9: 30-40% of MVC; Weeks 9-12: 40-50% of MVC; Weeks 12-18: sustain 50% of MVC. Incremental increases made at the 3, 6, 9, and 12-week clinic visits.
- Strength Walking w/ SRP: Home-Based Pedometer-Driven Walking Program plus SRP: Participants were given a pedometer to monitor daily steps and a weighted exercise vest at Week 7 to begin the strengthening component. A series of 10-minute lessons focused on increasing physical activity through lifestyle education and the use of a pedometer as a motivational tool.
  Participants maintain a daily training log. Pedometer readings used for setting activity goals. Initial step goals: 10% above the average 3-day pedometer step count at baseline. A 10% increase every other week, then a gradual increase when 30% above the baseline step count has been achieved. At week 7, participants will be given a vest to begin the strengthening component. The beginning weight load for the vest is calculated using 2% of baseline body weight and increased by the same amount every week until the end of the 12 weeks.
- NMES/Strength Walking w/ SRP: NMES, Home-Based Pedometer-Driven Walking Program plus SRP: This group will follow the protocol for both the NMES training and Strength Walking.
Period: Overall Study
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP
Started | 19 | 19 | 20 | 20
Completed | 13 | 11 | 11 | 15
Not Completed | 6 | 8 | 9 | 5
Not completed — Lost to Follow-up | 3 | 4 | 0 | 3
Not completed — Withdrawal by Subject | 3 | 4 | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP | Total
Number analyzed (Participants) | 19 | 19 | 20 | 20 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (8.4) | 35 (7.9) | 35 (11.3) | 33 (6.1) | 34 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 11 | 11 | 42
  Male | 9 | 9 | 9 | 9 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 8 | 11 | 8 | 13 | 40
  Race: African-American | 8 | 6 | 7 | 5 | 26
  Race: Asian/Pacific | 0 | 0 | 2 | 1 | 3
  Race: Multi-racial | 3 | 1 | 2 | 1 | 7
  Race: Missing | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Lower Extremity Muscle Strength- Extension
Description: Muscle strength was measured with a handheld dynamometer for extensor knee strength of the injured and uninjured knee.
Time Frame: 0, 3, 6, 9, 12, and 18 weeks
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP
Number analyzed (Participants) | 19 | 19 | 20 | 20
Kilograms
  Injured Knee: Week 0 | 27.5 (12.4) | 32.6 (14.7) | 32.1 (15.5) | 24.3 (11.4)
  Injured Knee: Week 3 | 25.4 (15.9) | 32 (10.4) | 30.4 (10.3) | 27.8 (13.7)
  Injured Knee: Week 6 | 23.3 (11.5) | 33.7 (11.5) | 29.8 (10) | 27.1 (13.4)
  Injured Knee: Week 9 | 26 (15.1) | 33.9 (13.6) | 29.2 (13.7) | 34 (16.8)
  Injured Knee: Week 12 | 27.8 (16) | 33 (10.6) | 32.7 (16.6) | 30.8 (14.8)
  Injured Knee: Week 18 | 28.5 (17.3) | 36.2 (10.2) | 31 (16.6) | 33.5 (15.8)
  Uninjured Knee: Week 0 | 28.2 (13) | 37.2 (16.4) | 36.2 (21.2) | 27.6 (14)
  Uninjured Knee: Week 3 | 26 (15.5) | 38.3 (18.8) | 34.5 (14.9) | 28 (13.8)
  Uninjured Knee: Week 6 | 25.4 (11.2) | 35.9 (13.9) | 34.2 (15.1) | 33.5 (19.4)
  Uninjured Knee: Week 9 | 27.2 (14) | 35.9 (15.1) | 29.8 (19.9) | 36.2 (18.3)
  Uninjured Knee: Week 12 | 25.8 (14.2) | 35.8 (12.6) | 33.8 (15.9) | 38.7 (22.6)
  Uninjured Knee: Week 18 | 27.6 (12) | 32.3 (9.1) | 33.2 (20.3) | 38.6 (22.1)

2. Primary Outcome: Lower Extremity Muscle Strength- Flexion
Description: Muscle strength was measured with a handheld dynamometer for flexor knee strength of the injured and uninjured knee.
Time Frame: 0, 3, 6, 9, 12, and 18 weeks
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP
Number analyzed (Participants) | 19 | 19 | 20 | 20
Kilograms
  Injured Knee: Week 0 | 16.2 (9.4) | 16.6 (7) | 16.2 (8.6) | 13.7 (6.9)
  Injured Knee: Week 3 | 15.3 (8.3) | 16.9 (4.8) | 17.8 (5.5) | 14.9 (7.4)
  Injured Knee: Week 6 | 15.4 (9.9) | 21.3 (12.1) | 15 (4.5) | 14.8 (5.9)
  Injured Knee: Week 9 | 15.6 (12.6) | 15.3 (4.9) | 15.9 (5.6) | 16.6 (7.2)
  Injured Knee: Week 12 | 14.5 (7.3) | 16.5 (4.5) | 18.4 (5.7) | 17.3 (7.4)
  Injured Knee: Week 18 | 14.7 (7.8) | 17.4 (4) | 15.4 (5.5) | 19.3 (10.4)
  Uninjured Knee: Week 0 | 20 (6.7) | 22.5 (8.4) | 22.6 (8) | 19.8 (8.6)
  Uninjured Knee: Week 3 | 20.1 (7.9) | 23.5 (8.2) | 22.7 (7.4) | 20.2 (7.5)
  Uninjured Knee: Week 6 | 16.9 (7.2) | 22.9 (6.6) | 19.8 (6.4) | 19.9 (10.3)
  Uninjured Knee: Week 9 | 17.5 (12.6) | 20.8 (5.2) | 23 (10.4) | 27.4 (15.7)
  Uninjured Knee: Week 12 | 17.3 (8.4) | 22.7 (6.4) | 25.9 (12.2) | 23 (11.1)
  Uninjured Knee: Week 18 | 18.1 (6.8) | 23.1 (8.2) | 24.1 (12) | 24.2 (11.3)

3. Primary Outcome: Lower Extremity Mobility- 6-Minute Walk Test
Description: Mobility was measured by the distance walked at a fast pace over 6-minutes,
Time Frame: 0, 6, 12, and 18 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP
Number analyzed (Participants) | 19 | 19 | 20 | 20
Inches
  Week 0 | 19800 (3398) | 20224 (5162) | 19728 (5347) | 18974 (4603)
  Week 6 | 21822 (4346) | 21696 (3905) | 22197 (3242) | 21696 (3905)
  Week 12 | 21404 (2534) | 22210 (3991) | 21595 (3092) | 20824 (6223)
  Week 18 | 21210 (3718) | 22984 (3390) | 22105 (3718) | 22945 (2883)

4. Primary Outcome: Lower Extremity Strength- Chair Test
Description: Mobility was measured by the number of complete standing and sitting cycles in 30-seconds
Time Frame: 0, 6, 12, and 18 weeks
Measure: Mean (Standard Deviation); unit: Rises
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP
Number analyzed (Participants) | 19 | 19 | 20 | 20
Rises
  Week 0 | 11.3 (3.7) | 11.4 (1.8) | 12.7 (3.9) | 10.7 (2.8)
  Week 6 | 12.7 (3.8) | 13.6 (2.6) | 14.4 (4) | 13.2 (1.9)
  Week 12 | 13.3 (4.8) | 13.9 (2.3) | 14.4 (2.3) | 14.5 (2.1)
  Week 18 | 13.3 (3.7) | 14.4 (1.5) | 15 (2.7) | 15.2 (2.2)

5. Primary Outcome: Lower Extremity Mobility and Endurance- Step Test
Description: Mobility and endurance were measured by the number of up and down step cycles completed in 2-minutes.
Time Frame: 0, 6, 12, and 18 weeks
Measure: Mean (Standard Deviation); unit: Step Cycles
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP
Number analyzed (Participants) | 19 | 19 | 20 | 20
Step Cycles
  Week 0 | 189 (67) | 162 (62) | 199 (60) | 172 (67)
  Week 6 | 185 (76) | 178 (78) | 224 (64) | 205 (75)
  Week 12 | 180 (82) | 235 (46) | 258 (42) | 202 (73)
  Week 18 | 202 (92) | 233 (75) | 224 (56) | 216 (73)

6. Secondary Outcome: Overall Pain Severity
Description: Pain severity was measured using item 3 from the IDKC Subjective Knee Evaluation: "If you have knee pain, how severe is it?" Participants responded using a scale of 0 (no pain) to 10 (worst pain imaginable). A mean pain score was calculated.
Time Frame: 0, 3, 6, 9, 12, and 18 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP
Number analyzed (Participants) | 19 | 19 | 20 | 20
score on a scale
  Week 0 | 5.4 (1.9) | 4.9 (2.1) | 5.7 (1.7) | 5.1 (1.9)
  Week 3 | 5.9 (2.3) | 5 (2.3) | 5.4 (1.9) | 5.0 (1.8)
  Week 6 | 6.2 (2.5) | 3.8 (1.6) | 5.3 (2.5) | 5.0 (2.3)
  Week 9 | 5.8 (2.4) | 4.1 (1.9) | 4.4 (1.7) | 4.3 (2.4)
  Week 12 | 5.3 (2.6) | 4.2 (2.1) | 5.1 (2.7) | 4.5 (2)
  Week 18 | 4.7 (3.1) | 3.6 (2.4) | 4.3 (2.4) | 3.9 (2.3)

7. Secondary Outcome: Knee Pain Following Performance Testing- 6-Minute Walk Test
Description: Knee pain intensity after the 6-Minute Walk Test was assessed using the Visual Analog Scale, an 11-point numerical rating scale. Participants rated current knee pain intensity on a scale of 0 (no pain) to 10 (worst pain imaginable). A mean pain score was calculated.
Time Frame: 0, 6, 12, and 18 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP
Number analyzed (Participants) | 19 | 19 | 20 | 20
score on a scale
  Week 0 | 2.4 (2.2) | 2.9 (2.4) | 1.8 (2.1) | 2.5 (2.1)
  Week 6 | 3.2 (2.5) | 1.6 (1.9) | 1.7 (2.8) | 1.4 (1.2)
  Week 12 | 2.7 (2.1) | 1.9 (2.1) | 1.6 (2.0) | 1.6 (1.7)
  Week 18 | 2.3 (2.1) | 1.6 (2.2) | 2.1 (2.9) | 1.2 (2.1)

8. Secondary Outcome: Knee Pain Following Performance Testing- Chair Stand Test
Description: Knee pain intensity after the 30-Second Chair Stand Test was assessed using the Visual Analog Scale, an 11-point numerical rating scale. Participants rated current knee pain intensity on a scale of 0 (no pain) to 10 (worst pain imaginable). A mean pain score was calculated.
Time Frame: 0, 6, 12, and 18 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP
Number analyzed (Participants) | 19 | 19 | 20 | 20
score on a scale
  Week 0 | 3.7 (2.3) | 2.5 (2.4) | 2.1 (1.9) | 2.7 (1.4)
  Week 6 | 3.5 (2.6) | 1.4 (1.8) | 1.4 (2.0) | 1.2 (1.4)
  Week 12 | 2.8 (2.2) | 2.0 (2.6) | 1.7 (2.5) | 1.2 (1.5)
  Week 18 | 2.4 (2.0) | 0.7 (0.9) | 1.5 (2.2) | 0.8 (1.5)

9. Secondary Outcome: Knee Pain Following Performance Testing- 2-Minute Step Test
Description: Knee pain intensity after the 2-Minute Step Test was assessed using the Visual Analog Scale, an 11-point numerical rating scale. Participants rated current knee pain intensity on a scale of 0 (no pain) to 10 (worst pain imaginable). A mean pain score was calculated.
Time Frame: 0, 6, 12, and 18 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP
Number analyzed (Participants) | 19 | 19 | 20 | 20
score on a scale
  Week 0 | 4.0 (2.4) | 3.7 (2.7) | 3.0 (2.1) | 3.7 (2.4)
  Week 6 | 3.5 (2.8) | 2.1 (2.5) | 2.5 (2.5) | 2.4 (1.4)
  Week 12 | 2.9 (2.6) | 3.0 (2.4) | 3.0 (2.4) | 1.9 (2.3)
  Week 18 | 2.6 (2.4) | 1.7 (2.4) | 2.1 (2.7) | 1.8 (2.6)

10. Secondary Outcome: Activities of Daily Living- Knee Symptoms
Description: The Activities of Daily Living Scale was used to measure self-perceived knee symptoms while performing typical activities. The knee symptom subscale ranges from "I do not have the symptom" to "The symptom prevents me from all daily activity". Scores ranged from 0-35. Higher scores are associated with diminished symptoms. A mean score was calculated.
Time Frame: 0, 3, 6, 9, 12, and 18 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP
Number analyzed (Participants) | 19 | 19 | 20 | 20
score on a scale
  Week 0 | 25.4 (4.7) | 23.3 (6.3) | 25.1 (5.2) | 22.9 (4.3)
  Week 3 | 25.0 (5.5) | 24.6 (6.9) | 26.2 (6.0) | 26 (2.8)
  Week 6 | 24.4 (6.5) | 27.9 (6.4) | 28.1 (4.7) | 27.4 (4.0)
  Week 9 | 25 (6.1) | 29.3 (6.6) | 29.6 (4.1) | 27.2 (4.7)
  Week 12 | 27.8 (6.3) | 26.5 (7.6) | 30.8 (3) | 27.6 (4.8)
  Week 18 | 29.6 (5.2) | 29.7 (4.7) | 30.9 (4.3) | 29.8 (4.7)

11. Secondary Outcome: Activities of Daily Living- Activity Limitation
Description: The Activities of Daily Living Scale was used to measure self-perceived limitations while performing typical activities. The limitation subscale ranges from "Activity is not difficult " to "I am unable to do the activity". Scores range from 0-45. Higher scores are associated with diminished symptoms. A mean score was calculated.
Time Frame: 0, 3, 6, 9, 12, and 18 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP
Number analyzed (Participants) | 19 | 19 | 20 | 20
score on a scale
  Week 0 | 32.9 (6.1) | 30.9 (4.9) | 30.9 (7.2) | 31.5 (2.4)
  Week 3 | 33.4 (6.4) | 33.3 (5.2) | 34.8 (5.8) | 33 (3.0)
  Week 6 | 33.5 (8.1) | 35.5 (5.5) | 34.9 (6.1) | 35.6 (4.4)
  Week 9 | 31.8 (6.9) | 39.8 (4.1) | 35.3 (5.8) | 36.5 (4.4)
  Week 12 | 32.9 (7.7) | 35.7 (5.9) | 36.7 (5.1) | 36.6 (5.4)
  Week 18 | 36.4 (6.7) | 38.1 (4.9) | 36.9 (6.0) | 38.6 (5.6)

ADVERSE EVENTS:
Arm/Group | Standard Rehabilitation Protocol (SRP) | NMES w/ SRP | Strength Walking w/ SRP | NMES/Strength Walking w/ SRP
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes